CLINICAL TRIAL: NCT07138950
Title: Hamstring Kasına UygulananStatik Germe ve Mulligan Bent Leg Raise Tekniğinin Fleksibilite ve Sıçrama Performansı Üzerine Akut Etkisi
Brief Title: Fexibility and Jump Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Tahir Keskin , Pt, PhD, Assistant Professor Tahir KESKİN, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: mulligan and jump performance
Record Dates: First submitted 2025-08-05; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hamstring Muscle Tightness; Static Stretching; Mulligan Mobilization; Jump Performance
MeSH Terms: interventions — Methods; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Arm 1 - Mulligan Grubu Arm Label: Mulligan
  Arm Type: Experimental
  Description: Participants receive Mulligan mobilization Arm 2 - stretching
  Arm Type: Experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BLR (Other)
  Interventions: Other: Mulligan Bent Leg Raise (BLR) Technique
- SS (Active Comparator)
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: Mulligan Bent Leg Raise (BLR) Technique — The Mulligan bent leg raise technique involves isometric contraction followed by stretches applied to the hamstring muscle in specific directions. The aim is to increase hamstring flexibility and active knee extension range of motion. The participant lay supine on an elevated bed, while the physiotherapist sat lateral to the leg to be stretched, placing the popliteal fossa of the participant's knee on their shoulder. The hip and knee of the leg to be stretched were flexed to 90°. Distraction was applied to the lower end of the femur, and the participant was asked to push the physiotherapist's shoulder with their leg and then relax. At this point of relaxation, the physiotherapist pushed the flexed knee as far forward as possible in the direction of hip flexion within a painless range. This position was held for 5 seconds at the end of the movement. Then, the neutral position was returned, and the procedure was repeated three times
  Arms: BLR
Other: Static Stretching — Participants lay supine on a stretcher with their backs straight. With the knee fully extended, the physical therapist placed the participant's leg on their shoulder and supported the ankle
  Arms: SS

SUMMARY:
This study was conducted to compare the effects of the static and Mulligan bent leg raise (BLR) techniques applied to address hamstring tightness on jumping performance. Participants with hamstring tightness participated in the study and were randomized into two groups. Group 1 (Classic Stretching Group) underwent a 30-second hamstring stretching protocol consisting of 5 repetitions. Participants in Group 2 underwent the BLR technique. Participants' active knee extension, vertical jump, and single-leg horizontal jump were measured before and after the study.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of hamstring muscle tightness.

Exclusion Criteria:

* Having any functional limitations that could affect test performance.
* Having any medical conditions that could affect the tests.
* Having more than 25° of limitation in the active knee extension test.
* Any lower extremity injury history within 2 years.
* Any neurological problem.
* Corticosteroid use.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
vertical jump | through study completion, an average of 5 months
Active Knee Extension Test | through study completion, an average of 5 months
one leg hop test | through study completion, an average of 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Üniversitesi Sağlık Bilimleri Fakültesi, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No